CLINICAL TRIAL: NCT03746262
Title: A Pilot Study of Changes in Circulating Tumor-Specific DNA (ctDNA) in Patients With Non-Metastatic Non-Small Cell Lung Cancer
Brief Title: Changes in Circulating Tumor-Specific DNA in Patients With Non-Metastatic Non-Small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Guardant Health, Inc. (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00036520; P30CA012197 (NIH); CCCWFU 62A15 (Other: NCI)
Record Dates: First submitted 2018-11-12; First posted 2018-11-19 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non-Metastatic Non-Small Cell Lung Cancer; Cancer; Lung Cancer; circulating tumor-specific DNA (ctDNA); non-invasive diagnostic
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood and tissue when available
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients - Stage I treated with surgery: ctDNA measures will be taken and descriptive statistics will be estimated. These include means, standard deviations, and 95% confidence intervals. Next, within group changes in ctDNA levels will be measured for each of the four groups. These change values will be estimated with 95% confidence intervals. In addition, paired t-tests will be performed to determine whether there were statistically significant changes in ctDNA levels at time points post-treatment or follow-up. After these paired analyses are performed, an exploratory longitudinal mixed model will be fit to examine the change in ctDNA levels.
- Patients - Stage I treated with radiotherapy: ctDNA measures will be taken and descriptive statistics will be estimated. These include means, standard deviations and 95% confidence intervals. Next, within group changes in ctDNA levels will be measured for each of the four groups. These change values will be estimated with 95% confidence intervals. In addition, paired t-tests will be performed to determine whether there were statistically significant changes in ctDNA levels at time points post-treatment or follow-up. After these paired analyses are performed, an exploratory longitudinal mixed model will be fit to examine the change in ctDNA levels.
- Patients - Stage II treated with surgery & chemotherapy: ctDNA measures will be taken and descriptive statistics will be estimated. These include means, standard deviations and 95% confidence intervals. Next, within group changes in ctDNA levels will be measured for each of the four groups. These change values will be estimated with 95% confidence intervals. In addition, paired t-tests will be performed to determine whether there were statistically significant changes in ctDNA levels at time points post-treatment or follow-up. After these paired analyses are performed, an exploratory longitudinal mixed model will be fit to examine the change in ctDNA levels.
- Patients - Stage III treated with chemoradiotherapy: ctDNA measures will be taken and descriptive statistics will be estimated. These include means, standard deviations and 95% confidence intervals. Next, within group changes in ctDNA levels will be measured for each of the four groups. These change values will be estimated with 95% confidence intervals. In addition, paired t-tests will be performed to determine whether there were statistically significant changes in ctDNA levels at time points post-treatment or follow-up. After these paired analyses are performed, an exploratory longitudinal mixed model will be fit to examine the change in ctDNA levels.

SUMMARY:
The purpose of this research study is to evaluate a blood test to measure circulating tumor DNA (ctDNA). It is hypothesized that ctDNA may identify patients who can be considered for additional therapy. 40 People with non-metastatic non-small cell lung cancer will be asked to take part in this study. Participants will have approximately 3 teaspoons of blood withdrawn from a vein at three different times. These times will be before primary treatment (either surgery or radiation therapy), 1 month after primary treatment, and 4 months after primary treatment.

DETAILED DESCRIPTION:
The purpose of this research study is to evaluate a blood test to measure circulating tumor DNA (ctDNA). It is hypothesized that ctDNA may identify patients who can be considered for additional therapy. 40 People with non-metastatic non-small cell lung cancer will be asked to take part in this study. Participants will have approximately 3 teaspoons of blood withdrawn from a vein at three different times. These times will be before primary treatment (either surgery or radiation therapy), 1 month after primary treatment, and 4 months after primary treatment. The total amount of blood withdrawn during the study will be approximately 9 teaspoons. Participants will be followed every 3 months for 12 months to determine if a confirmed recurrence or progression has occurred. Participants will also be asked to complete questionnaires on their quality of life and their smoking behaviors. As part of this study, a blood sample will be obtained and DNA from participants blood sample will be purified. DNA, or deoxyribonucleic acid, stores and transmits inherited traits, such as eye color or blood type. As part of this research project, participant's DNA will be studied in an effort to find out if there are genes that contribute to medical conditions like their cancer that are part of the study. If participants have surgery to have tumor removed or if participants have a biopsy of their tumor, the study would like to take some of the leftover tissue to purify and study the DNA from the tissue sample.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed or clinically suspected stage I, II or III NSCLC, provided such patients will be scheduled for a procedure that will provide histologic confirmation of the diagnosis (if the procedure does not provide histologic confirmation of the diagnosis of NSCLC the particular patient will be removed from the study and replaced).
* Scheduled for treatment with surgery or radiotherapy (Stage I), surgery and chemotherapy (Stage II), or chemoradiotherapy (Stage III). For stage I receiving radiotherapy, treatment must be stereotactic body radiation therapy (SBRT) consisting of 3-5 fractions.
* Ability to provide blood sample at the following time points: pre-treatment, 1 month post definitive treatment, and 4 post definitive treatment.
* Ability to understand and the willingness to sign an IRB-approved informed consent document.
* Staging studies including PET-CT for all patients prior to the initiation of primary treatment, as a pretreatment requirement. For patients with Stage II and III, MRI or CT of the brain is needed prior to the initiation of primary treatment. Patients, however, may be registered and have the pretreatment blood sample collected, provided that the staging studies are being scheduled. Registered patients who are found, after screening tests, to have Stage IV disease will be removed from the study and replaced.

Exclusion Criteria:

* Females who are pregnant
* History of organ transplant.
* For stage II and III patients, must be able to receive chemotherapy.
* Active cardiovascular issues in the past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women of all races and ethnicities who meet the above-described eligibility criteria are eligible to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-05-13 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2018-08-10 (Actual)

PRIMARY OUTCOMES:
Change in ctDNA levels in patients with Stage I or II (Non-small cell lung cancer) NSCLC | up to 12 months
  ctDNA levels in patients with Stage I or II NSCLC treated with surgery compared with ctDNA levels in the rest of the cohort. Comparisons will be made at the following time points: Pre-treatment, Post-treatment, and Follow-up.
Change in ctDNA levels in patients with Stage III NSCLC | up to 12 months
  ctDNA levels in patients with Stage III NSCLC treated with chemoradiotherapy compared with ctDNA levels in the rest of the cohort. Comparisons will be made at the following time points: Pre-treatment, Post-treatment , and Follow-up.
Change in ctDNA by treatment group | up to 12 months
  To determine the change in ctDNA by treatment group at the following time points: change from Pre-treatment to Post-treatment, and change from Pre-treatment to Follow-up.

SECONDARY OUTCOMES:
Health Related Quality of Life- (HRQL) | up to 12 months
  A two part questionnaire, will be used to assess HRQL: (1) QLQ-C30, a core questionnaire covering general aspects of HRQL, and (2) QLQ-LC13, a lung cancer specific questionnaire. For the QLQ-C30 - All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. For the QLQ-LC13 - All of the scales and single-item measures range in score from 0 to 100. A high score for the scales and single items represents a high level of symptomatology or problems.
Number of Packs Smoked Per Day | up to 12 months
  The number of packs of tobacco participants smoked per day will be assessed and recorded
Number of Years Smoked | up to 12 months
  The number of years participants smoked will be recorded.
Number of Participants that have a Smoking Status | up to 12 months
  Participants will be asked about their current smoking status (yes/no). These answers will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Grant, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anker P, Mulcahy H, Chen XQ, Stroun M. Detection of circulating tumour DNA in the blood (plasma/serum) of cancer patients. Cancer Metastasis Rev. 1999;18(1):65-73. doi: 10.1023/a:1006260319913. PMID 10505546
- [Background] Sorenson GD, Pribish DM, Valone FH, Memoli VA, Bzik DJ, Yao SL. Soluble normal and mutated DNA sequences from single-copy genes in human blood. Cancer Epidemiol Biomarkers Prev. 1994 Jan-Feb;3(1):67-71. PMID 8118388
- [Background] Minamoto T, Yamashita N, Ochiai A, Mai M, Sugimura T, Ronai Z, Esumi H. Mutant K-ras in apparently normal mucosa of colorectal cancer patients. Its potential as a biomarker of colorectal tumorigenesis. Cancer. 1995 Mar 15;75(6 Suppl):1520-6. doi: 10.1002/1097-0142(19950315)75:6+3.0.co;2-l. PMID 7889485
- [Background] Sorenson GD. Detection of mutated KRAS2 sequences as tumor markers in plasma/serum of patients with gastrointestinal cancer. Clin Cancer Res. 2000 Jun;6(6):2129-37. PMID 10873061
- [Background] Sorenson GD. A review of studies on the detection of mutated KRAS2 sequences as tumor markers in plasma/serum of patients with gastrointestinal cancer. Ann N Y Acad Sci. 2000 Apr;906:13-6. doi: 10.1111/j.1749-6632.2000.tb06582.x. No abstract available. PMID 10818588
- [Background] Kirk GD, Camus-Randon AM, Mendy M, Goedert JJ, Merle P, Trepo C, Brechot C, Hainaut P, Montesano R. Ser-249 p53 mutations in plasma DNA of patients with hepatocellular carcinoma from The Gambia. J Natl Cancer Inst. 2000 Jan 19;92(2):148-53. doi: 10.1093/jnci/92.2.148. PMID 10639517
- [Background] Jackson PE, Qian GS, Friesen MD, Zhu YR, Lu P, Wang JB, Wu Y, Kensler TW, Vogelstein B, Groopman JD. Specific p53 mutations detected in plasma and tumors of hepatocellular carcinoma patients by electrospray ionization mass spectrometry. Cancer Res. 2001 Jan 1;61(1):33-5. PMID 11196182
- [Background] Shao ZM, Wu J, Shen ZZ, Nguyen M. p53 mutation in plasma DNA and its prognostic value in breast cancer patients. Clin Cancer Res. 2001 Aug;7(8):2222-7. PMID 11489795 (Retraction: PMID 12231550 Shao ZM, Wu J, Shen ZZ, Nguyen M. Clin Cancer Res. 2002 Sep;8(9):3027)
- [Background] Silva JM, Gonzalez R, Dominguez G, Garcia JM, Espana P, Bonilla F. TP53 gene mutations in plasma DNA of cancer patients. Genes Chromosomes Cancer. 1999 Feb;24(2):160-1. PMID 9885984
- [Background] Mayall F, Jacobson G, Wilkins R, Chang B. Mutations of p53 gene can be detected in the plasma of patients with large bowel carcinoma. J Clin Pathol. 1998 Aug;51(8):611-3. doi: 10.1136/jcp.51.8.611. PMID 9828821
- [Background] Bruhn N, Beinert T, Oehm C, Jandrig B, Petersen I, Chen XQ, Possinger K, Fleischhacker M. Detection of microsatellite alterations in the DNA isolated from tumor cells and from plasma DNA of patients with lung cancer. Ann N Y Acad Sci. 2000 Apr;906:72-82. doi: 10.1111/j.1749-6632.2000.tb06594.x. PMID 10818600
- [Background] Chen XQ, Stroun M, Magnenat JL, Nicod LP, Kurt AM, Lyautey J, Lederrey C, Anker P. Microsatellite alterations in plasma DNA of small cell lung cancer patients. Nat Med. 1996 Sep;2(9):1033-5. doi: 10.1038/nm0996-1033. PMID 8782463
- [Background] Gonzalez R, Silva JM, Sanchez A, Dominguez G, Garcia JM, Chen XQ, Stroun M, Provencio M, Espana P, Anker P, Bonilla F. Microsatellite alterations and TP53 mutations in plasma DNA of small-cell lung cancer patients: follow-up study and prognostic significance. Ann Oncol. 2000 Sep;11(9):1097-104. doi: 10.1023/a:1008305412635. PMID 11061602
- [Background] Nawroz H, Koch W, Anker P, Stroun M, Sidransky D. Microsatellite alterations in serum DNA of head and neck cancer patients. Nat Med. 1996 Sep;2(9):1035-7. doi: 10.1038/nm0996-1035. PMID 8782464
- [Background] Taback B, Giuliano AE, Hansen NM, Hoon DS. Microsatellite alterations detected in the serum of early stage breast cancer patients. Ann N Y Acad Sci. 2001 Sep;945:22-30. doi: 10.1111/j.1749-6632.2001.tb03860.x. PMID 11708482
- [Background] Taback B, O'Day SJ, Boasberg PD, Shu S, Fournier P, Elashoff R, Wang HJ, Hoon DS. Circulating DNA microsatellites: molecular determinants of response to biochemotherapy in patients with metastatic melanoma. J Natl Cancer Inst. 2004 Jan 21;96(2):152-6. doi: 10.1093/jnci/djh011. PMID 14734706
- [Background] Taback B, Fujiwara Y, Wang HJ, Foshag LJ, Morton DL, Hoon DS. Prognostic significance of circulating microsatellite markers in the plasma of melanoma patients. Cancer Res. 2001 Aug 1;61(15):5723-6. PMID 11479206
- [Background] Goessl C, Heicappell R, Munker R, Anker P, Stroun M, Krause H, Muller M, Miller K. Microsatellite analysis of plasma DNA from patients with clear cell renal carcinoma. Cancer Res. 1998 Oct 15;58(20):4728-32. PMID 9788629
- [Background] Muller HM, Widschwendter M. Methylated DNA as a possible screening marker for neoplastic disease in several body fluids. Expert Rev Mol Diagn. 2003 Jul;3(4):443-58. doi: 10.1586/14737159.3.4.443. PMID 12877384
- [Background] Collisson E, Mortimer S, Sebisanovic D, et al. Biopsy-free comprehensive tumor profiling of 1,000+ consecutive cancer patients using CLIA-certified commercial test and its clinical utility. Paper presented at: 2015 AACR Annual Meeting. Abstract #2403. 2015.
- [Background] Talasaz A, Mortimer S, Sebisanovic D, et al. Use of the GUARDANT360 noninvasive tumor sequencing assay on 300 patients across colorectal, melanoma, lung, breast, and prostate cancers and its clinical utility. J Clin Oncol 32, 2014 (suppl; abstr e22041).
- [Background] Austin LK, Avery T, Jaslow R, et al. Concordance of circulating tumor DNA (ctDNA) and next-generation sequencing (NGS) as molecular monitoring tools in metastatic breast cancer (MBC). Paper presented at: 2015 AACR Annual Meeting. Abstract #4918. 2015.
- [Background] Austin LK, Jaslow R, Avery T, et al. Clinical utility of circulating tumor DNA (ctDNA) in advanced and metastatic breast cancer. Paper presented at: 2015 AACR Annual Meeting. Abstract #4928. 2015.
- [Background] Piccioni DE, Lanman RB, Nagy RJ, Talasaz A, Pingle SC, Kesari S. Analysis of cell-free circulating tumor DNA in patients with glioblastoma and other primary brain tumors. Paper presented at: 2015 ASCO Annual Meeting. J Clin Oncol 33, 2015 (suppl; abstr 11072). 2015.
- [Background] Heatherton TF, Kozlowski LT, Frecker RC, Fagerstrom KO. The Fagerstrom Test for Nicotine Dependence: a revision of the Fagerstrom Tolerance Questionnaire. Br J Addict. 1991 Sep;86(9):1119-27. doi: 10.1111/j.1360-0443.1991.tb01879.x. PMID 1932883